CLINICAL TRIAL: NCT05291078
Title: Exploring the Effects of Transcutaneous Trigeminal Nerve Stimulation Using NUEYNE-T30 and NUEYNE-T100 and Sound Fusion Stimulation on Tinnitus: A Single-center, Double Blind, Placebo-controlled Group, Investigator Initiated Study (IIT) Study
Brief Title: Study of Application of Transcutaneous Trigeminal Nerve Stimulation and Sound Fusion Stimulation on Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nu Eyne Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NE_TNT_IIT001
Record Dates: First submitted 2022-03-08; First posted 2022-03-22 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2022-03

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group A (Experimental): Tinnitus patients(n=12 people)
  Interventions: Device: A transcutaneous trigeminal nerve stimulator: High Frequency; Device: Sound Therapy
- Experimental Group B (Experimental): Tinnitus patients(n=12 people)
  Interventions: Device: A transcutaneous trigeminal nerve stimulator: Low Frequency; Device: Sound Therapy
- Control Group (Sham Comparator): Tinnitus patients(n=12 people)
  Interventions: Device: A transcutaneous trigeminal nerve stimulator: Sham; Device: Sound Therapy

INTERVENTIONS:
Device: A transcutaneous trigeminal nerve stimulator: High Frequency — 30min/day, at least 5 to 7 times a week
  Arms: Experimental Group A
Device: A transcutaneous trigeminal nerve stimulator: Low Frequency — 30min/day, at least 5 to 7 times a week
  Arms: Experimental Group B
Device: A transcutaneous trigeminal nerve stimulator: Sham — 30min/day, at least 5 to 7 times a week
  Arms: Control Group
Device: Sound Therapy — Notch Therapy at least 30min/day, at least 5 to 7 times a week

SUMMARY:
This study aims to evaluate the efficacy of applying transcutaneous trigeminal nerve stimulation (NUEYNE-T30, NUEYNE-T100) and sound fusion stimulation on tinnitus.

DETAILED DESCRIPTION:
Duration of study period (per participant): Screening period (-7~0 days), Intervention period (30 days) Patient needs to visit site at least 3 times (Screening, V1, V2). V1 can be done with screening visit. Tele-visit should be done on day 15.

ELIGIBILITY:
Inclusion Criteria:

* adults suffering from tinnitus
* Participants must be 19 to 70 years of age, at the time of screening
* Patient who suffers from tinnitus symptom more than 3 months and scores more than 18(criteria of mild) in Tinnitus Handicap Inventory (THI) examination
* Patients with a hearing threshold of 70dB or less when calculated using the quadrant method in the pure tone audiometry
* A person who has no physical or mental restrictions in participating in clinical trial
* Those who voluntarily agreed to participate in clinical trials
* A person who has no pregnancy plan and has agreed to the contraceptive plan for infertile women during the intervention period of clinical trial

Exclusion Criteria:

* A person who does not meet the inclusion criteria
* A person who has difficulty communicating and conducting examinations.
* The disease of the outer or middle ear or central nervous system.
* Subjects who have difficulty conducting clinical trials due to intellectual or cognitive impairment
* Pregnant or lactating women
* A person who cannot understand or read ICF (illiterate or foreigner)
* A person who received tinnitus treatment (blood circulation enhancer, tranquilizer, tinnitus masker, biofeedback etc.) within 2 weeks of baseline or plans to receive it.
* A person who is difficult to participate in a clinical trial according to the researcher's judgment. (e.g., heart-related problems, seizure, epilepsy. Patients transplanted metal or electronic device in head & neck. Patient suffering from unknown pain. Patients who are warned not to use out clinical trial device or is prohibited from using it.)

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Changes in Tinnitus handicap inventory(THI) score | baseline, 4 weeks
  Check the changes in Tinnitus handicap inventory(THI) score
  The score on the questionnaire ranges from 0 to 100. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Changes in Loudness of Tinnitogram | baseline, 4 weeks
  Check the changes in Loudness of Tinnitogram
Changes in Minimal masking level of Tinnitogram | baseline, 4 weeks
  Check the changes in Minimal masking level of Tinnitogram
Changes in Tinnitus magnitude index(TMI) score | baseline, 4 weeks
  Check the changes in Tinnitus magnitude index(TMI) score
  The questionnaire consists of three questions. The score for No. 1 question ranges from 0 to 10. The score for No. 2 question ranges from 0% to 10%. The score for No. 2 question ranges from 0mm to 100mm. Higher scores mean a worse outcome.
Changes in EEG | baseline, 4 weeks
  Check the changes in EEG
Changes in PPG | baseline, 4 weeks
  Check the changes in PPG
Changes in Beck Depression Inventory(BDI) score | baseline, 4 weeks
  Check the changes in Beck Depression Inventory score
  The score on the questionnaire ranges from 0 to 63. Higher scores mean a worse outcome.
Changes in Pittsburg Sleep Quality Index (PSQI) score | baseline, 4 weeks
  Check the changes in Pittsburg Sleep Quality Index (PSQI) score
  The score on the questionnaire ranges from 0 to 21. Higher scores mean a worse outcome.
Changes in MOS Short-Form 36-Item Health Survey(SF-36) score | baseline, 4 weeks
  Check the changes in MOS Short-Form 36-Item Health Survey(SF-36) score
  The questionnaire consists of 8 subscales. The score for each subscale ranges from 0 to 100. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Iljoon Moon, Ph. D., MD., Principal Investigator — Department of Otorhinolaryngology, Samsung Medical Center
Locations (1):
- Department of Otorhinolaryngology, Samsung Medical Center, Seoul, South Korea